CLINICAL TRIAL: NCT03095209
Title: Observation Study of Patients With Non-Small Cell Lung Cancer and Esophageal Cancer Treated With Chemo-Radiation Followed by Surgery
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: RT-103
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Lung Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Standard of care concurrent chemo-radiation therapy
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks (maximum 12 weeks post-CRT) after finishing CRT with surgical aspects determined by the treating surgical oncologist.
Drug: Paclitaxel — chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks (maximum 12 weeks post-CRT) after finishing CRT with surgical aspects determined by the treating surgical oncologist.
Radiation: Radiation Therapy — The total radiation dose will be 50.4 Gy in daily fraction of 1.8 Gy for esophageal cancer and 60 Gy in daily fraction of 2 Gy for non-small cell lung cancer.

SUMMARY:
Patients on this observation study must have planned treatment regimen with concurrent CRT followed by planned surgery, which is considered as standard of care for their disease. The total radiation dose will be 50.4 Gy in daily fraction of 1.8 Gy for esophageal cancer and 60 Gy in daily fraction of 2 Gy for non-small cell lung cancer. The concurrent chemo regimen will carboplatin-paclitaxel managed by the treating medical oncologist. Patients are planned to receive surgery at approximately 6 to 9 weeks (maximum 12 weeks post-CRT) after finishing CRT with surgical aspects determined by the treating surgical oncologist.

Patients on this observation study will donate their blood samples within 4 weeks before initiating CRT, within 1 week before completing CRT, 1 month after CRT, and 1 month after surgery (or 3 months after CRT if surgery is not done for any reason). They are also requested to fill out questionnaires (EORTC QLQ-30, EORTC QLQ-OES18, and Pain Scale as attached) prior to CRT, weekly during CRT, 1 month after CRT, 1 month after surgery (or 3 months after CRT if surgery is not done for any reason), and 6 months after CRT. Any patients with incomplete treatment will have samples collected up to the point where they discontinue. The specimen collection, handling and processing will be done by Protocol Support Lab (PSL) at Fox Chase Cancer Center under the directions of the Director, R. Katherine Alpaugh, PhD, following the procedures outlined in PSL lab manual. The patients in this observation study will be asked to donate a tissue specimen after the definitive surgery for investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have pathologically-confirmed and previously untreated:

   * Non-small cell lung cancer, Stage IIIA (T1-3 N2 M0); OR
   * Localized esophageal cancer, ≥T2, or N+, and M0 according to the American Joint Committee on Cancer (AJCC) 7th edition staging.
2. The planned treatment regimen must be concurrent chemoradiation with Carboplatin-Paclitaxel followed by surgery.
3. Age > 18 years.
4. ECOG performance status is 0-1.
5. Laboratory studies must meet each of the following criteria (with labs drawn within 4 weeks prior to the registration):

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   * Platelets ≥100,000 cells/mm3
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable)
   * Creatinine ≤2 X the upper limit of normal
   * Bilirubin ≤ 1.5 X upper limit of normal
   * AST ≤ 3 X upper limit of normal
6. Men and women of childbearing potential must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy completed.
7. Patients must be able to read and write English to comply with the questionnaire portions of the protocol.
8. Subjects must sign a written informed study consent and HIPAA consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.

Exclusion Criteria:

1. Patients who have had previous radiotherapy in the thorax.
2. Patients who have a history of ataxia telangiectasia or other documented history of radiation hypersensitivity.
3. Patients who have a history scleroderma or other active connective tissue disease.

9 Women of childbearing potential must not be pregnant and non-lactating. They are required to have a negative serum pregnancy test within 72 hours prior to registration or they can decline the pregnancy test with the specific supporting reason such as not sexually active or using birth control; postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential; woman status post oophorectomy or hysterectomy are considered non-childbearing potential.

4 Patients who have uncontrolled inter-current illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for the phase I trial (RT-101) but decline to enroll should be offered to participate in this parallel observation study. Patients with the following disease will be included in this observation study:
  I. non-small cell lung cancer, Stage IIIA (T1-3 N2 M0) II. localized esophageal cancer, ≥T2, or N+, and M0
  Patients on this observation study must have planned treatment regimen with concurrent CRT followed by planned surgery, which is considered as standard of care for their disease.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Serum inflammation markers | 7 months
  Serum inflammation markers will be analyzed that will serve as the control for the parallel study RT-101. In the 7 month period the blood will be drawn once during the following months - 1, 2,3, 7

SECONDARY OUTCOMES:
Quality of life and pain | 1 year
  Quality of life will be assessed in the form of surveys which reveal the ability to complete daily activities the pain level of the patient. During the study the surveys will be conducted in the following months- month1, month 2 (every week that is 4 times), month 3, month 7 and month 9. If there are delays due to toxicities the survey collection timelines can shift and the last survey could be collected up to 12 months. The number of surveys collected will be the same.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No